CLINICAL TRIAL: NCT04318184
Title: First Exercise Reports of Diabetes Centre: Effects of Exercise on Metabolic Parameters in Patients With Type 2 Diabetes Mellitus
Brief Title: Effects of Exercise on Metabolic Parameters in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17073117-050.06
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise; Type-2 Diabetes Mellitus treatment; Body Composition; Blood Samples; Blood Pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Submaximal aerobic exercise protocol
  Interventions: Procedure: Aerobic exercise

INTERVENTIONS:
Procedure: Aerobic exercise — The aerobic exercise protocol was performed 3 times a week for 3 months on the treadmill. Loading periods were performed according to the heart rate maximum using the Karvonen formula (%60-80 Heart rate maximum)

SUMMARY:
Diabetes is considered an epidemic disease with the 463 million affected patients (between 20-79 years) and it is estimated that 578 million people will have diabetes by 2030 [1]. According to The International Diabetes Federation (IDF) reports, 4,2 million adults were considered to die due to diabetes and its complications in 2019. Because of this situation, diabetes treatment is so important. The recommendations for the treatment of DM include medications and lifestyle management, which includes physical activity (PA), medical nutrition therapy, smoking cessation counseling, and psychosocial care. PA is an important aspect of management that directly under the control of the patients. So the investigators want to interrogate the effect of exercise on blood parameters, blood pressure, body compositions.

DETAILED DESCRIPTION:
The data of the participants who came to the sports center where is prepared for the diabetes patients in the hospital will be collected from the past registration files on the electronic system.

Sociodemographic data, blood values and bio-impedance measurements of each patient are collected coming to the sports center, routinely.

Patients who had missing data, patients who did not complete the 3-month exercise program were excluded from the analysis. All analyses were performed using the Statistical Package for the Social Sciences (SPSS) version 22. 0 for Windows. Data are expressed as mean ± standard deviation. The one-sample Kolmogorov-Smirnov test was performed to assess the distribution of data. Due to their distribution, numerical variables in different subjects were compared with the t-test or Mann-Whitney U test. Comparison of variables before and after the exercise program were compared by the paired t-test (parametric variable) or Wilcoxon test (non-parametric variable). Probability values were two-tailed, and a p-value of less than 0.05 was considered as significant.

All assessments were performed in the clinic at baseline and end of the 3rd month. The blood samples were collected. The systolic and diastolic blood pressure (SBP and DBP) were measured with an automatic arm BP monitor before and after every session. Body mass and body composition, including percent body fat, fat and fat-free mass, were determined using a bioelectric impedance system with the electrodes in contact with soles and heels of both feet. At the baseline and end of the third month, the same person repeated all assessments.

Patients had recruited 3 sessions a week for 3 months (Monday/Wednesday/Friday). Every session consisted of aerobic exercise protocol and warm-up, cooldown period. Patients aerobic loading capacity was calculated before the every session using by Karvonen formula as submaximal loading.

ELIGIBILITY:
Inclusion Criteria:

1. Persons who were diagnosed with DM,
2. Aged between 18 and 65 years,
3. Patients who completed the three-month exercise program.

Exclusion Criteria:

1. Had chronic drug (antidiabetic and antilipidemic) adjustments for 3 months at the beginning and during the exercise program,
2. Participated in an exercise program before,
3. Had a health condition other than DM associated with glucose metabolism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
"Change" is being assessed for HbA1c | Baseline and end of the 3rd month
  Blood parameters
"Change" is being assessed Total Cholesterol | Baseline and end of the 3rd month
  Blood parameters
"Change" is being assessed for LDL | Baseline and end of the 3rd month
  Blood parameters
"Change" is being assessed for HDL | Baseline and end of the 3rd month
  Blood parameters
"Change" is being assessed for Blood Glucose | Baseline and end of the 3rd month
  Blood parameters
"Change" is being assessed for Post prandial glucose | Baseline and end of the 3rd month
  Blood parameters
"Change" is being assessed for Triglyceride | Baseline and end of the 3rd month
  Blood parameters

SECONDARY OUTCOMES:
"Change" is being assessed for Blood Pressure | Baseline and end of the 3rd month
  Sistolic and Diastolic Pressure
"Change" is being assessed for Fat Mass (kg) | Baseline and end of the 3rd month
  Evaluation with bio-empedans device (TANITA)
"Change" is being assessed for Muscle Mass (kg) | Baseline and end of the 3rd month
  Evaluation with bio-empedans device (TANITA)
"Change" is being assessed for BMI | Baseline and end of the 3rd month
  Evaluation with bio-empedans device (TANITA)

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No